## 知情同意书

项目名称:天津市糖尿病视网膜病变社区筛查研究 方案版本号及版本日期:01,2024年1月29日 知情同意书版本号及版本日期:01,2024年1月29日 亲爱的居民(受试者):

您好!我们将邀请您参加《天津市糖尿病视网膜病变筛查项目》,本知情同意书将提供给您一些信息以帮助您决定是否参加本项目,您参加本项目是自愿的。如果您有意愿加入本项目,请看下列说明。项目目的:

我们希望通过临床检查和问卷调查两部分内容了解天津市糖尿病视网膜病变的患病率及其影响因素,提升基层医疗卫生机构糖尿病患者并发症发现干预能力,构建上下联动的糖尿病防治网络;坚持预防为主、防治结合的工作方针,探索适宜我市的糖尿病防控模式;广泛开展宣传教育,提升患者自我管理意识,提高糖尿病视网膜病变筛查率,降低致盲率。

## 具体内容:

如果您同意参与本项目,我们将对每位受试者进行编号,建立病 历档案,您将接受如下检查:

临床检查包括:空腹抽血,视力、验光和眼底照相等眼科检查,其中 眼底相机将搭载眼科智能影像管理系统(云平台),获得的眼底相片 将在保证信息隐私的前提下使用 AI 与眼科医师相结合的形式进行阅 片。在研究过程中我们需要采集一些您的标本,将由专业人员为您取 样,例如从您的胳膊上抽取静脉血 10 毫升,留取尿液 10 毫升,共需 1 次。其中,5ml 由检验科工作人员进行血常规与血生化检测,剩余 5ml 样本储存于我院生物样本库,可能用于未来眼科相关疾病的科学 研究。部分复合适应症的患者还将接受下肢血管彩色多普勒超声,中 医四诊合参检查和经络检查。

问卷调查包括:基本信息、内科疾病、视觉质量问卷、生活质量、眼科症状与疾病、药物史、疾病家族史、女性专有题目等。

## 风险与受益

风险:①您在检查过程中,眼部可能存在一定的风险或不适,如一过性视物模糊等。②必要时需要对您的瞳孔进行散瞳处理,其风险与标准散瞳检查一样。如果需要进行散瞳处理,我们将使用眼保健医生常规使用的散瞳药物。有些人可能会对散瞳药物有过敏反应,为了减少风险,医生将提前询问患者是否有青光眼或其它眼部疾病,以及是否对此类散瞳药物有过敏或其它不适的反应。③空腹抽血可能导致低血糖、低血压甚至晕厥。另外标本的采集可能会有一些非常小的风险,包括短暂的疼痛、局部青紫,少数人会有轻度头晕,或极为罕见的针头感染。

受益:①参加调查的受试者可以免费获得一份详细的眼科检查报告。②如有需要进一步诊疗的眼部疾病,可开通绿色通道,及时给予治疗。

## 隐私问题:

如果您决定参加本项目,您参加试验及在试验中的个人资料均属

保密。对于您来说,所有的信息将是保密的,除非获得您的许可,否则可以识别您身份的信息将不会透露给项目小组以外的成员。所有的项目成员和项目申办方都被要求对您的身份保密。您的档案仅供项目人员查阅,但为确保项目按照规定进行,必要时,政府管理部门或伦理审查委员会的成员可以按规定在项目单位查阅您的个人资料。希望能够得到您的支持与帮助!

(由调查员询问后填写)

知情同意签字:

我已经阅读了本知情同意书,并且我的医生\_\_\_\_\_(签字)已经将此项目的目的、内容、风险和受益情况向我作了详细的解释说明,对我询问的所有问题也给予了解答,我对此项目已经了解,我自愿参加本项目。

筛查对象签名: 年 月

调查员签名: 年 月 日

(注:如果受试者不识字时尚需见证人签名,如果受试者无行为能力时则需代理人同意)

Н